CLINICAL TRIAL: NCT03605589
Title: A Pilot Study of Blinatumomab in Combination With a PD1 Inhibitor, Pembrolizumab, in Pediatric and Young Adult Patients With Relapsed/Refractory CD19 Positive B-cell Acute Leukemia or Lymphoma
Brief Title: Pembro + Blina Combination in Pediatric and Young Adult Patients With Relapsed/Refractory Acute Leukemia or Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment due to the availability of other novel salvage therapies for relapsed/refractory B-ALL.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pembro-EB-1701
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Leukemia, B-cell; Lymphoma, B-Cell
Keywords: Blinatumomab; Pembrolizumab; CD19 positive; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Recurrence | interventions — blinatumomab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a pilot study to assess the safety, tolerability, and preliminary anti-tumor activity of the combination of pembrolizumab and blinatumomab in children and young adult patients with relapsed and/or refractory CD19 positive B-cell hematologic malignancies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab and Pembrolizumab (Experimental): Blinatumomab and Pembrolizumab will be given for 2 cycles (each cycle lasts 35 days).
  Blinatumomab administered as a continuous IV infusion. Patient Weight Greater Than or Equal to 45 kg (Fixed dose) Patient Weight Less Than 45 kg (BSA-based dose)
  Cycle 1 (Days 1-7):
  Patient Weight Greater Than or Equal to 45 kg: 9 mcg/day Patient Weight Less Than 45 kg: 5 mcg/m2/day
  Cycle 1(Days 8-28):
  Patient Weight Greater Than or Equal to 45 kg: 28 mcg/day Patient Weight Less Than 45 kg: 15 mcg/m2/day
  Cycle 2 (Days 1-28):
  Patient Weight Greater Than or Equal to 45 kg: 28 mcg/day Patient Weight Less Than 45 kg: 15 mcg/m2/day
  Pembrolizumab: 2 mg/kg (max dose 200 mg) administered as a 30 minute IV infusion on day 12 of cycle 1 and day 5 of cycle 2.
  Interventions: Drug: Blinatumomab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Blinatumomab — Continuous IV infusion
  Other Names: Blincyto
Drug: Pembrolizumab — IV infusion
  Other Names: Keytruda

SUMMARY:
This study combines the immune checkpoint inhibitor pembrolizumab with the BITE antibody blinatumomab for the treatment of relapsed/refractory pre-B cell ALL. Pembrolizumab at the proposed dosing schedule has been very well tolerated in adult studies, including elderly and unfit patients, as well as in pediatric patients. Both blinatumomab and pembrolizumab are FDA-approved for use in children as well as adults. Phase I/II trials in adult patients have demonstrated safety and activity of pembrolizumab in combination with multiple agents. In this trial, the combination of pembrolizumab and blinatumomab will be investigated for toxicity as well as possible synergy in the treatment of relapsed/refractory pre-B cell ALL.

This is a single institution investigator-initiated pilot study designed to test the safety and feasibility of combining pembrolizumab and blinatumomab immunotherapies in children, adolescents, and young adults with CD19 positive hematologic malignancies. The investigator will define the toxicity profile of the combination in two safety strata based on whether or not a patient has had a prior allogeneic hematopoietic stem cell transplant (HSCT), as they hypothesize that the immune toxicities may differ between strata. In addition, the overall response rate (CR/CRh) to this therapy will be estimated. Additional biologic correlates will be conducted to delineate the effect of the combination therapy on the patient's leukemia/lymphoma and T-cell populations and how this may influence response to therapy.

DETAILED DESCRIPTION:
Participants who meet study eligibility will receive or continue to receive blinatumomab by continuous IV infusion for 28 days and also receive pembrolizumab (by IV infusion over 30 minutes) on day 12 of cycle 1 and day 5 of cycle 2.

One cycle lasts 35 days and patients will receive 2 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-40
* Diagnosis of CD19 positive B-cell acute lymphoblastic leukemia (ALL) positive B-cell acute lymphoblastic leukemia (ALL) or CD19 positive B-cell lymphoma
* Patients with CD19 positive B-ALL must have greater than or equal to 5% lymphoblast in the bone marrow AND meet one of the following criteria:
* 2nd or greater relapse
* Any relapse after allo-HSCT
* Refractory disease
* Patients with CD19 positive relapsed/refractory lymphoma must be in 2nd or greater relapse or have refractory disease with the markers of disease burden
* Patients with CNS 1 or CNS 2 leukemia are eligible.Patients with CNS 3 leukemia are not eligible. However, patients with a history of CNS 3 status who have been sufficiently treated are eligible if currently CNS 1 or 2. Patients with an isolated CNS relapse are not eligible.
* Karnofsky performance level greater than or equal to 50 % for patients older than 16
* Lansky performance level greater than or equal to 50 % less than or equal to 16
* Patients recovered from acute toxicities from prior anti-cancer chemotherapy including HSCT, cytotoxic therapy, prior blinatumomab, biologic, immunotherapy, monoclonal antibody, XRT and corticosteroid therapy
* Patients with adequate hematological, renal, liver, cardiac, pulmonary and CNS organ functions
* Female participants of child bearing age must have negative pregnancy test, abstain or use contraception for 120 days after last dose of pembrolizumab

Exclusion Criteria:

* Patients with the following diagnoses: CNS 3 leukemia, CNS lymphoma, active GVHD, Downs Syndrome, CNS or testicular relapse, optic nerve or retinal involvement requiring radiation therapy
* Pregnant or breastfeeding
* Concomitant corticosteroids, immunosuppressive therapies, investigational drugs, anti-cancer agents
* Concurrent illnesses including: history of any grade autoimmune disorder, Grade 2 or higher hypothyroidism die to autoimmunity, uncontrolled infection, interstitial lung disease or pneumonitis
* Patients with other concurrent malignancies
* Patients who have received live vaccines within the last 30 days
* Patients with history of solid organ transplant

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of combining pembrolizumab and blinatumomab (dose limiting toxicities) | 2 cycles of therapy (70 days)
  Number of DLTs
Treatment related toxicities | 2 cycles of therapy (70 days)
  Number of related adverse events

SECONDARY OUTCOMES:
Disease response | 2 cycles (70 days)
  Estimate of overall response rate (CR/CRh)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Breese, MD. PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escherich G, Horstmann MA, Zimmermann M, Janka-Schaub GE; COALL study group. Cooperative study group for childhood acute lymphoblastic leukaemia (COALL): long-term results of trials 82,85,89,92 and 97. Leukemia. 2010 Feb;24(2):298-308. doi: 10.1038/leu.2009.249. Epub 2009 Dec 17. PMID 20016530
- [Background] Moricke A, Zimmermann M, Reiter A, Henze G, Schrauder A, Gadner H, Ludwig WD, Ritter J, Harbott J, Mann G, Klingebiel T, Zintl F, Niemeyer C, Kremens B, Niggli F, Niethammer D, Welte K, Stanulla M, Odenwald E, Riehm H, Schrappe M. Long-term results of five consecutive trials in childhood acute lymphoblastic leukemia performed by the ALL-BFM study group from 1981 to 2000. Leukemia. 2010 Feb;24(2):265-84. doi: 10.1038/leu.2009.257. Epub 2009 Dec 10. PMID 20010625
- [Background] Schmiegelow K, Forestier E, Hellebostad M, Heyman M, Kristinsson J, Soderhall S, Taskinen M; Nordic Society of Paediatric Haematology and Oncology. Long-term results of NOPHO ALL-92 and ALL-2000 studies of childhood acute lymphoblastic leukemia. Leukemia. 2010 Feb;24(2):345-54. doi: 10.1038/leu.2009.251. Epub 2009 Dec 10. PMID 20010622
- [Background] Stary J, Zimmermann M, Campbell M, Castillo L, Dibar E, Donska S, Gonzalez A, Izraeli S, Janic D, Jazbec J, Konja J, Kaiserova E, Kowalczyk J, Kovacs G, Li CK, Magyarosy E, Popa A, Stark B, Jabali Y, Trka J, Hrusak O, Riehm H, Masera G, Schrappe M. Intensive chemotherapy for childhood acute lymphoblastic leukemia: results of the randomized intercontinental trial ALL IC-BFM 2002. J Clin Oncol. 2014 Jan 20;32(3):174-84. doi: 10.1200/JCO.2013.48.6522. Epub 2013 Dec 16. PMID 24344215
- [Background] Gaynon PS. Childhood acute lymphoblastic leukaemia and relapse. Br J Haematol. 2005 Dec;131(5):579-87. doi: 10.1111/j.1365-2141.2005.05773.x. PMID 16351633
- [Background] Raetz EA, Bhatla T. Where do we stand in the treatment of relapsed acute lymphoblastic leukemia? Hematology Am Soc Hematol Educ Program. 2012;2012:129-36. doi: 10.1182/asheducation-2012.1.129. PMID 23233571
- [Background] Tallen G, Ratei R, Mann G, Kaspers G, Niggli F, Karachunsky A, Ebell W, Escherich G, Schrappe M, Klingebiel T, Fengler R, Henze G, von Stackelberg A. Long-term outcome in children with relapsed acute lymphoblastic leukemia after time-point and site-of-relapse stratification and intensified short-course multidrug chemotherapy: results of trial ALL-REZ BFM 90. J Clin Oncol. 2010 May 10;28(14):2339-47. doi: 10.1200/JCO.2009.25.1983. Epub 2010 Apr 12. PMID 20385996
- [Background] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Background] von Stackelberg A, Locatelli F, Zugmaier G, Handgretinger R, Trippett TM, Rizzari C, Bader P, O'Brien MM, Brethon B, Bhojwani D, Schlegel PG, Borkhardt A, Rheingold SR, Cooper TM, Zwaan CM, Barnette P, Messina C, Michel G, DuBois SG, Hu K, Zhu M, Whitlock JA, Gore L. Phase I/Phase II Study of Blinatumomab in Pediatric Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2016 Dec 20;34(36):4381-4389. doi: 10.1200/JCO.2016.67.3301. Epub 2016 Oct 31. PMID 27998223
- [Background] Kantarjian HM, Stein AS, Bargou RC, Grande Garcia C, Larson RA, Stelljes M, Gokbuget N, Zugmaier G, Benjamin JE, Zhang A, Jia C, Topp MS. Blinatumomab treatment of older adults with relapsed/refractory B-precursor acute lymphoblastic leukemia: Results from 2 phase 2 studies. Cancer. 2016 Jul 15;122(14):2178-85. doi: 10.1002/cncr.30031. Epub 2016 May 3. PMID 27143254
- [Background] Talmadge JE, Donkor M, Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. Cancer Metastasis Rev. 2007 Dec;26(3-4):373-400. doi: 10.1007/s10555-007-9072-0. PMID 17717638
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Chen L, Zincke H, Blute ML, Leibovich BC, Kwon ED. Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. Cancer. 2005 Nov 15;104(10):2084-91. doi: 10.1002/cncr.21470. PMID 16208700
- [Background] McDermott DF, Atkins MB. PD-1 as a potential target in cancer therapy. Cancer Med. 2013 Oct;2(5):662-73. doi: 10.1002/cam4.106. Epub 2013 Jul 21. PMID 24403232
- [Background] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Background] Muro K, Chung HC, Shankaran V, Geva R, Catenacci D, Gupta S, Eder JP, Golan T, Le DT, Burtness B, McRee AJ, Lin CC, Pathiraja K, Lunceford J, Emancipator K, Juco J, Koshiji M, Bang YJ. Pembrolizumab for patients with PD-L1-positive advanced gastric cancer (KEYNOTE-012): a multicentre, open-label, phase 1b trial. Lancet Oncol. 2016 Jun;17(6):717-726. doi: 10.1016/S1470-2045(16)00175-3. Epub 2016 May 3. PMID 27157491
- [Background] Plimack ER, Bellmunt J, Gupta S, Berger R, Chow LQ, Juco J, Lunceford J, Saraf S, Perini RF, O'Donnell PH. Safety and activity of pembrolizumab in patients with locally advanced or metastatic urothelial cancer (KEYNOTE-012): a non-randomised, open-label, phase 1b study. Lancet Oncol. 2017 Feb;18(2):212-220. doi: 10.1016/S1470-2045(17)30007-4. Epub 2017 Jan 10. PMID 28081914
- [Background] Nanda R, Chow LQ, Dees EC, Berger R, Gupta S, Geva R, Pusztai L, Pathiraja K, Aktan G, Cheng JD, Karantza V, Buisseret L. Pembrolizumab in Patients With Advanced Triple-Negative Breast Cancer: Phase Ib KEYNOTE-012 Study. J Clin Oncol. 2016 Jul 20;34(21):2460-7. doi: 10.1200/JCO.2015.64.8931. Epub 2016 May 2. PMID 27138582
- [Background] Armand P, Shipp MA, Ribrag V, Michot JM, Zinzani PL, Kuruvilla J, Snyder ES, Ricart AD, Balakumaran A, Rose S, Moskowitz CH. Programmed Death-1 Blockade With Pembrolizumab in Patients With Classical Hodgkin Lymphoma After Brentuximab Vedotin Failure. J Clin Oncol. 2016 Nov 1;34(31):3733-3739. doi: 10.1200/JCO.2016.67.3467. PMID 27354476
- [Background] Costa R, Carneiro BA, Agulnik M, Rademaker AW, Pai SG, Villaflor VM, Cristofanilli M, Sosman JA, Giles FJ. Toxicity profile of approved anti-PD-1 monoclonal antibodies in solid tumors: a systematic review and meta-analysis of randomized clinical trials. Oncotarget. 2017 Jan 31;8(5):8910-8920. doi: 10.18632/oncotarget.13315. PMID 27852042
- [Background] Kong Y, Zhang J, Claxton DF, Ehmann WC, Rybka WB, Zhu L, Zeng H, Schell TD, Zheng H. PD-1(hi)TIM-3(+) T cells associate with and predict leukemia relapse in AML patients post allogeneic stem cell transplantation. Blood Cancer J. 2015 Jul 31;5(7):e330. doi: 10.1038/bcj.2015.58. PMID 26230954
- [Background] Wherry EJ, Kurachi M. Molecular and cellular insights into T cell exhaustion. Nat Rev Immunol. 2015 Aug;15(8):486-99. doi: 10.1038/nri3862. PMID 26205583
- [Background] Zhou Q, Munger ME, Veenstra RG, Weigel BJ, Hirashima M, Munn DH, Murphy WJ, Azuma M, Anderson AC, Kuchroo VK, Blazar BR. Coexpression of Tim-3 and PD-1 identifies a CD8+ T-cell exhaustion phenotype in mice with disseminated acute myelogenous leukemia. Blood. 2011 Apr 28;117(17):4501-10. doi: 10.1182/blood-2010-10-310425. Epub 2011 Mar 8. PMID 21385853
- [Background] Feucht J, Kayser S, Gorodezki D, Hamieh M, Doring M, Blaeschke F, Schlegel P, Bosmuller H, Quintanilla-Fend L, Ebinger M, Lang P, Handgretinger R, Feuchtinger T. T-cell responses against CD19+ pediatric acute lymphoblastic leukemia mediated by bispecific T-cell engager (BiTE) are regulated contrarily by PD-L1 and CD80/CD86 on leukemic blasts. Oncotarget. 2016 Nov 22;7(47):76902-76919. doi: 10.18632/oncotarget.12357. PMID 27708227
- [Background] McClanahan F, Hanna B, Miller S, Clear AJ, Lichter P, Gribben JG, Seiffert M. PD-L1 checkpoint blockade prevents immune dysfunction and leukemia development in a mouse model of chronic lymphocytic leukemia. Blood. 2015 Jul 9;126(2):203-11. doi: 10.1182/blood-2015-01-622936. Epub 2015 Mar 23. PMID 25800048
- [Background] Armand P, Nagler A, Weller EA, Devine SM, Avigan DE, Chen YB, Kaminski MS, Holland HK, Winter JN, Mason JR, Fay JW, Rizzieri DA, Hosing CM, Ball ED, Uberti JP, Lazarus HM, Mapara MY, Gregory SA, Timmerman JM, Andorsky D, Or R, Waller EK, Rotem-Yehudar R, Gordon LI. Disabling immune tolerance by programmed death-1 blockade with pidilizumab after autologous hematopoietic stem-cell transplantation for diffuse large B-cell lymphoma: results of an international phase II trial. J Clin Oncol. 2013 Nov 20;31(33):4199-206. doi: 10.1200/JCO.2012.48.3685. Epub 2013 Oct 14. PMID 24127452
- [Background] Carbognin L, Pilotto S, Milella M, Vaccaro V, Brunelli M, Calio A, Cuppone F, Sperduti I, Giannarelli D, Chilosi M, Bronte V, Scarpa A, Bria E, Tortora G. Differential Activity of Nivolumab, Pembrolizumab and MPDL3280A according to the Tumor Expression of Programmed Death-Ligand-1 (PD-L1): Sensitivity Analysis of Trials in Melanoma, Lung and Genitourinary Cancers. PLoS One. 2015 Jun 18;10(6):e0130142. doi: 10.1371/journal.pone.0130142. eCollection 2015. PMID 26086854
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Background] Topp MS, Gokbuget N, Zugmaier G, Klappers P, Stelljes M, Neumann S, Viardot A, Marks R, Diedrich H, Faul C, Reichle A, Horst HA, Bruggemann M, Wessiepe D, Holland C, Alekar S, Mergen N, Einsele H, Hoelzer D, Bargou RC. Phase II trial of the anti-CD19 bispecific T cell-engager blinatumomab shows hematologic and molecular remissions in patients with relapsed or refractory B-precursor acute lymphoblastic leukemia. J Clin Oncol. 2014 Dec 20;32(36):4134-40. doi: 10.1200/JCO.2014.56.3247. Epub 2014 Nov 10. PMID 25385737
- [Background] Kohnke T, Krupka C, Tischer J, Knosel T, Subklewe M. Increase of PD-L1 expressing B-precursor ALL cells in a patient resistant to the CD19/CD3-bispecific T cell engager antibody blinatumomab. J Hematol Oncol. 2015 Oct 8;8:111. doi: 10.1186/s13045-015-0213-6. PMID 26449653
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Foran AE, Nadel HR, Lee AF, Savage KJ, Deyell RJ. Nivolumab in the Treatment of Refractory Pediatric Hodgkin Lymphoma. J Pediatr Hematol Oncol. 2017 Jul;39(5):e263-e266. doi: 10.1097/MPH.0000000000000703. PMID 27841828
- [Background] Davids MS, Kim HT, Bachireddy P, Costello C, Liguori R, Savell A, Lukez AP, Avigan D, Chen YB, McSweeney P, LeBoeuf NR, Rooney MS, Bowden M, Zhou CW, Granter SR, Hornick JL, Rodig SJ, Hirakawa M, Severgnini M, Hodi FS, Wu CJ, Ho VT, Cutler C, Koreth J, Alyea EP, Antin JH, Armand P, Streicher H, Ball ED, Ritz J, Bashey A, Soiffer RJ; Leukemia and Lymphoma Society Blood Cancer Research Partnership. Ipilimumab for Patients with Relapse after Allogeneic Transplantation. N Engl J Med. 2016 Jul 14;375(2):143-53. doi: 10.1056/NEJMoa1601202. PMID 27410923
- [Background] Onizuka M, Kojima M, Matsui K, Machida S, Toyosaki M, Aoyama Y, Kawai H, Amaki J, Hara R, Ichiki A, Ogawa Y, Kawada H, Nakamura N, Ando K. Successful treatment with low-dose nivolumab in refractory Hodgkin lymphoma after allogeneic stem cell transplantation. Int J Hematol. 2017 Jul;106(1):141-145. doi: 10.1007/s12185-017-2181-9. Epub 2017 Jan 17. PMID 28097534
- [Background] Shad AT, Huo JS, Darcy C, Abu-Ghosh A, Esposito G, Holuba MJ, Robey N, Cooke KR, Symons HJ, Chen AR, Llosa NJ. Tolerance and effectiveness of nivolumab after pediatric T-cell replete, haploidentical, bone marrow transplantation: A case report. Pediatr Blood Cancer. 2017 Mar;64(3). doi: 10.1002/pbc.26257. Epub 2016 Sep 21. PMID 27650634
- [Background] Villasboas JC, Ansell SM, Witzig TE. Targeting the PD-1 pathway in patients with relapsed classic Hodgkin lymphoma following allogeneic stem cell transplant is safe and effective. Oncotarget. 2016 Mar 15;7(11):13260-13264. doi: 10.18632/oncotarget.7177. PMID 26848626
- [Background] Yared JA, Hardy N, Singh Z, Hajj S, Badros AZ, Kocoglu M, Yanovich S, Sausville EA, Ujjani C, Ruehle K, Goecke C, Landau M, Rapoport AP. Major clinical response to nivolumab in relapsed/refractory Hodgkin lymphoma after allogeneic stem cell transplantation. Bone Marrow Transplant. 2016 Jun;51(6):850-2. doi: 10.1038/bmt.2015.346. Epub 2016 Feb 1. No abstract available. PMID 26828905
- [Background] Haverkos BM, Abbott D, Hamadani M, Armand P, Flowers ME, Merryman R, Kamdar M, Kanate AS, Saad A, Mehta A, Ganguly S, Fenske TS, Hari P, Lowsky R, Andritsos L, Jagasia M, Bashey A, Brown S, Bachanova V, Stephens D, Mineishi S, Nakamura R, Chen YB, Blazar BR, Gutman J, Devine SM. PD-1 blockade for relapsed lymphoma post-allogeneic hematopoietic cell transplant: high response rate but frequent GVHD. Blood. 2017 Jul 13;130(2):221-228. doi: 10.1182/blood-2017-01-761346. Epub 2017 May 3. PMID 28468799
- [Background] Patel SP, Kurzrock R. PD-L1 Expression as a Predictive Biomarker in Cancer Immunotherapy. Mol Cancer Ther. 2015 Apr;14(4):847-56. doi: 10.1158/1535-7163.MCT-14-0983. Epub 2015 Feb 18. PMID 25695955
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Routh JC, Ashley RA, Sebo TJ, Lohse CM, Husmann DA, Kramer SA, Kwon ED. B7-H1 expression in Wilms tumor: correlation with tumor biology and disease recurrence. J Urol. 2008 May;179(5):1954-9; discussion 1959-60. doi: 10.1016/j.juro.2008.01.056. Epub 2008 Mar 20. PMID 18355839
- [Background] Topp MS, Gokbuget N, Zugmaier G, Degenhard E, Goebeler ME, Klinger M, Neumann SA, Horst HA, Raff T, Viardot A, Stelljes M, Schaich M, Kohne-Volland R, Bruggemann M, Ottmann OG, Burmeister T, Baeuerle PA, Nagorsen D, Schmidt M, Einsele H, Riethmuller G, Kneba M, Hoelzer D, Kufer P, Bargou RC. Long-term follow-up of hematologic relapse-free survival in a phase 2 study of blinatumomab in patients with MRD in B-lineage ALL. Blood. 2012 Dec 20;120(26):5185-7. doi: 10.1182/blood-2012-07-441030. Epub 2012 Sep 28. PMID 23024237
- [Background] Poschke I, Flossdorf M, Offringa R. Next-generation TCR sequencing - a tool to understand T-cell infiltration in human cancers. J Pathol. 2016 Dec;240(4):384-386. doi: 10.1002/path.4800. Epub 2016 Oct 21. PMID 27569598
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Background] Harris AC, Young R, Devine S, Hogan WJ, Ayuk F, Bunworasate U, Chanswangphuwana C, Efebera YA, Holler E, Litzow M, Ordemann R, Qayed M, Renteria AS, Reshef R, Wolfl M, Chen YB, Goldstein S, Jagasia M, Locatelli F, Mielke S, Porter D, Schechter T, Shekhovtsova Z, Ferrara JL, Levine JE. International, Multicenter Standardization of Acute Graft-versus-Host Disease Clinical Data Collection: A Report from the Mount Sinai Acute GVHD International Consortium. Biol Blood Marrow Transplant. 2016 Jan;22(1):4-10. doi: 10.1016/j.bbmt.2015.09.001. Epub 2015 Sep 16. PMID 26386318
- [Background] Paczesny S, Hakim FT, Pidala J, Cooke KR, Lathrop J, Griffith LM, Hansen J, Jagasia M, Miklos D, Pavletic S, Parkman R, Russek-Cohen E, Flowers ME, Lee S, Martin P, Vogelsang G, Walton M, Schultz KR. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: III. The 2014 Biomarker Working Group Report. Biol Blood Marrow Transplant. 2015 May;21(5):780-92. doi: 10.1016/j.bbmt.2015.01.003. Epub 2015 Jan 30. PMID 25644957